CLINICAL TRIAL: NCT02677376
Title: Validation of Imaging-Based Biomarkers of Treatment Response in Patients With Metastatic Castration-Resistant Prostate Cancer Treated With Enzalutamide
Brief Title: Imaging Biomarkers to Validate Response in Enzalutamide-Treated mCRPC
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UW15052; 2015-1174 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2016-01-08; First posted 2016-02-09 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: 18F-Sodium Fluoride (NaF) — NaF is a tracer (dye) that will show changes to the cancer in bones. By using this tracer with PET/CT imaging, our ability to evaluate and measure changes in bone lesions could be greatly improved. Participants will have a NaF PET/CT scan within 14 days prior to starting enzalutamide. All subjects will undergo a second NaF PET/CT scan after taking enzalutamide for 12 weeks. The NaF PET/CT obtained at week 12 will be compared to the first NaF PET/CT to identify a bone tumor that is responding (shrinking) and a bone tumor that is not responding (not shrinking).

SUMMARY:
To determine the feasibility and success rate of tumor tissue procurement using molecular-image-directed biopsies of responding and non-responding osseous metastases, measured by NaF PET/CT, in patients with metastatic castrate-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate.
* Identifiable prostate cancer-related osseous metastases on bone scan or NaF PET/CT in the vertebral body, pelvis or other bone. Such lesions must be amenable to serial NaF PET/CT imaging. Preference will be given to subjects with multiple lesions that can be imaged in one image acquisition session to obtain maximal information as well as locations of lesions amenable to bone biopsies.
* Patients must be starting enzalutamide for treatment of metastatic castrate-resistant prostate, with cycle 1 day 1 occurring within 14 days after the first baseline NaF PET/CT. Subjects will be allowed to receive enzalutamide treatment on a concurrent study as long as the enzalutamide treatment study does not prohibit concurrent participation.
* Men of all races and ethnic groups of age ≥18 years.
* The effects of NaF on the developing human fetus are unknown. For this reason and because radiopharmaceuticals used for diagnostic imaging and other therapeutic agents and imaging procedures used in this trial may be or are known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Patients must be able to comply with all study procedures, including having both the ability and willingness to lie flat for ≥ 30 minutes during imaging and undergo bone biopsies.
* Patients must have both the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known bleeding diathesis or on therapeutic anticoagulants (warfarin, low-molecular heparin, heparin analogues) that would increase risk of complications from bone biopsies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sodium fluoride F-18 (NaF).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men ≥18 years with progressive, bone-metastatic castrate-resistant prostate cancer who will be treated with enzalutamide will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
The percentage of biopsies obtained from NaF PET/CT- identified responding and non-responding bone metastases that contain tumor tissue from 30 patients | 12 weeks
  To determine the feasibility and success rate of tumor tissue procurement using molecular-image-directed biopsies of responding and non-responding osseous metastases, measured by NaF PET/CT, in patients with metastatic castrate-resistant prostate cancer.

SECONDARY OUTCOMES:
The number of known response molecular biomarkers obtained from responding lesions as identified using NaF PET/CT in 30 patients who have received 12 weeks of enzalutamide. | Within 2 weeks of week 12
  To compare NaF PET/CT responding lesions to known response molecular biomarkers obtained from biopsy of responding lesions
The number of patients whose biopsy tissue demonstrates at least 5 markers from a panel of 300 individual markers that have a moderate effect size of 1.0 or greater for the difference between the enzalutamide resistant and responding bone metastases | Within 2 weeks of week 12
  To compare NaF PET/CT non-responding lesions to known resistance molecular biomarkers obtained from biopsy of non-responding lesions
Characterizations obtained from NaF PET/CT images from patients who demonstrate a progression free survival of greater than 12 months on enzalutamide treatment. | Within 2 weeks of week 12
  To determine NaF PET/CT -derived radiomic profiles that correlate with prolonged benefit (PFS > 12 month) to enzalutamide
Comparison of the percentage of responding/non-responding lesions on NaF PET/CT to PSA response, RECIST response, time to PSA progressions and radiographic progression free survival | Within 2 weeks of week 12
  To correlate global responsiveness on NaF PET/CT (percentage of responding/non-responding lesions, SUVtotal) with clinical outcomes: PSA response, RECIST response, time to PSA progressions, and radiographic PFS

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, Principal Investigator — Principal Investigator
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/